CLINICAL TRIAL: NCT03339102
Title: Post-marketing Surveillance Study of Adalimumab (Humira®) for Non-infectious Intermediate, Posterior, or Panuveitis Patients According to the Standard for "Re-examination of New Drugs"
Brief Title: Post-marketing Surveillance Study of Adalimumab (Humira®) for Non-infectious Intermediate, Posterior, or Panuveitis Patients
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P17-176
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Non-infectious Intermediate, Posterior and Panuveitis
Keywords: Non-infectious intermediate, posterior and panuveitis; Post-Marketing Surveillance; Humira®
MeSH Terms: conditions — Panuveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants who received Humira®: Non-infectious intermediate, posterior, or panuveitis patients who received Humira®

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Humira® (Adalimumab) for the treatment of non-infectious intermediate, posterior, or panuveitis patients under a routine treatment practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with Non-infectious intermediate, posterior and pan-uveitis
* Patients voluntarily signed a patient authorization & informed consent form.
* Decision on the treatment with Humira® was made prior to any decision to approach the patient to participate in this study.
* Humira® treatment is indicated as per local Summary of Product Characteristics (SmPC) and professional and/or reimbursement guidelines.

Exclusion Criteria:

* A patient who are contraindications to originator adalimumab (Humira®) as listed on the approved Korean label.
* A patient who is participating on other interventional clinical trials
* Prior treatment with Humira®, including current course of Humira® started prior to baseline visit assessments.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-infectious intermediate, posterior and panuveitis (NIIPPU) patients who had been prescribed with Humira® will be registered to the study in accordance with the drug approval status as well as the investigator's clinical judgment.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of patients reported with serious adverse event | Up to Week 32
  The patients reported with serious adverse event will be collected.

SECONDARY OUTCOMES:
Change in Visual acuity | Up to follow-up week 22
  The change in visual acuity is assessed from the best corrected visual acuity achieved after the first dose on visual acuity chart in each eye.
Assessing Presence /absence of new active inflammatory chorioretinal lesions | Up to follow-up week 22
  Presence or absence of new active inflammatory chorioretinal lesions is assessed.
Assessing Treatment Response | Up to follow-up week 22
  Treatment response is assessed as improvement, no improvement and aggravation.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (17):
- South Korea (17):
  - Pusan National University Hosp /ID# 202026, Busan, Busan Gwang Yeogsi
  - Soon Chun Hyang University Cheonan Hospital /ID# 204551, Cheonan, Chungcheongnam-do
  - Yeungnam University Med Ctr /ID# 201361, Daegu, Daegu Gwang Yeogsi
  - Seoul National Univ Bundang ho /ID# 201657, Seongnam, Gyeonggido
  - Ajou University Hospital /ID# 201516, Suwon, Gyeonggido
  - HanGil Eye Hospital /ID# 201655, Bupyeong, Incheon Gwang Yeogsi
  - Wonkwang University Hospital /ID# 204545, Iksan, Jeonrabugdo
  - Nune Eye Hospital /ID# 211613, Seoul, Seoul
  - Gangnam Severance Hospital /ID# 202027, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 201515, Seoul, Seoul Teugbyeolsi
  - Maryknoll Medical Center /ID# 201370, Busan
  - Chungbuk National Univ Hosp /ID# 204544, Cheongju-si
  - Apgujung St. Mary's Eye Center /ID# 210721, Gangnam-gu
  - Inje University Ilsan Paik Hos /ID# 204543, Goyang
  - Chosun University Hospital /ID# 204542, Gwangju
  - Seoul National University Hospital /ID# 201656, Seoul
  - Kim's Eye Hospital /ID# 205685, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/adalimumab_P17-176.pdf